CLINICAL TRIAL: NCT03964935
Title: The Effect of Lycopene Antioxidant Gel Compared to Minocycline Hydrochloride Microspheres as Adjunctive to Non Surgical Periodontal Treatment by Measuring Matrix Metalloproteinase-9, Transforming Growth Factor-Beta 1, Interleukin-8, and Tissue Inhibitor of Metalloproteinases -1
Brief Title: Lycopene vs Minocycline Hydrochloride as Adjunctive to Periodontal Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Ali A Abdulkareem, Lecturer, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 013618
Record Dates: First submitted 2019-05-20; First posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Periodontal Pocket
MeSH Terms: conditions — Periodontal Pocket | interventions — Lycopene; Minocycline; Powders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lycopene (Experimental): Prepared by solving lycopene powder in a solvent (ethanol: propylene glycol: water in the ratio of 50:30:20). The solution was then gelled by adding 8% hydroxypropyl cellulose (HPC). The concentration of the prepared gel equals to 2%.
  After scaling, root planing, and polishing (SRP), the gel delivered into periodontal pocket using insulin syringes, the therapeutic dose is about 2mg/0.1 ml.
  Interventions: Drug: Lycopene
- Minocycline HCL (Active Comparator): Minocycline HCL Microspheres, 1mg minocycline powder per cartridge. A locally applied antibiotic that is placed directly into the infected periodontal pocket following SCR.
  Interventions: Drug: Minocycline HCl 1mg Oral Powder
- Distilled water (Placebo Comparator): Used to irrigate periodontal pockets after SRP
  Interventions: Other: Distilled water

INTERVENTIONS:
Drug: Lycopene — Prepared by solving lycopene powder in a solvent (ethanol: propylene glycol: water in the ratio of 50:30:20). The solution was then gelled by adding 8% hydroxypropyl cellulose (HPC). The concentration of the prepared gel equals to 2%.
  After SRP, the gel delivered into periodontal pocket using insulin syringes, the therapeutic dose is about 2mg/0.1 ml.
  Arms: Lycopene
Drug: Minocycline HCl 1mg Oral Powder — Minocycline HCl Microspheres, 1mg minocycline powder per cartridge. A locally applied antibiotic that is placed directly into the infected periodontal pocket following SCR.
  Arms: Minocycline HCL
Other: Distilled water — Used to irrigate periodontal pockets after SRP
  Arms: Distilled water

SUMMARY:
Periodontal diseases are among the most common medical conditions that may influence humans; 50% of the adult population can be affected by this illness. The condition is usually initiated by lack or reduction in oral hygiene which is then aggravated by the presence of microorganisms within biofilm which will induce a sequel of events that will lead to periodontitis. Scaling, root planning, and polishing (SRP) are the golden standard procedures in the treatment. Systemic antibiotics as adjunctive therapy has been established to be an excellent modality in controlling the bacterial virulence, hence, supporting the conventional SRP therapy. in order to avoid and limit the harmful effect of systemic antibiotics different locally applied preparations have been introduced including antioxidants. The aim of this prospective clinical study is to compare between the effect of Minocycline hydrochloride (HCL) microsphere and Lycopene gel when they are applied intrapocket subgingival with conventional SRP therapy

DETAILED DESCRIPTION:
Periodontal diseases are among the most common medical conditions that may influence humans; 50% of the adult population can be affected by this illness. The condition is usually initiated by lack or reduction in oral hygiene which is then aggravated by the presence of microorganisms within biofilm which will induce a sequel of events that will lead to periodontitis. The multifactorial nature of the disease necessitates a multifactorial approach to restore the balance within the oral echo system. Scaling, root planning, and polishing (SRP) are the golden standard procedures in the treatment; the therapeutic nature of these clinical intervention is based on disrupting the biofilm and stimulate the host defense mechanism to have the upper hand in targeting the microorganisms and their toxins. Systemic antibiotics as adjunctive therapy has been established to be an excellent modality in controlling the bacterial virulence, hence, supporting the conventional SRP therapy; in order to avoid and limit the harmful effect of systemic antibiotics different locally applied preparations have been introduced. Clinical parameters bleeding on probing (BOP), pocket depth (PD), and clinical attachment level (CAL) have been improved when Minocycline hydrochloride (HCL) microspheres was locally applied as an adjunctive drug to conventional SRP. Oxidative stress is another factor related to periodontitis. The free radicals are a by-product of the inflammatory reaction induced by the disease progression; free radicals eliminated by antioxidants which is naturally found in the diet especially fruits and vegetables; however, when the imbalance occur and the free radicals over weighed the antioxidants there will be further initiation of the destruction mechanism. The role of antioxidant as therapeutic agent in reducing the oxidative stress has been well studied and their supporting effect to the conventional SRP treatment is well documented. Lycopene extract can be applied as a gel intrapocket subgingival and it can have a promising result with the SRP.

The aim of this prospective clinical study is to compare between the effect of Minocycline HCL microsphere and Lycopene gel when they are applied intrapocket subgingival with conventional SRP therapy. The study will utilize split mouth technique; three sites within the oral cavity that have a pocket depth greater than 5 mm will be included. Each site will be designated to receive a specific treatment, Control group (site) will have SRP and water irrigation treatment, active group (site) will have local application of Minocycline HCL gel following SRP therapy, and the experimental site which will receive lycopene and SRP treatment. The influence of these therapeutic agents will be determined by the expression of selected inflammation-related markers in the gingival crevicular fluid collected from the experimental sites. The markers that will be examined are MMP-9, interleukin (IL)-8, TGF-Beta 1, and TIMP1. The change in the clinical parameters will be measured before the commencement of treatment and it will be examined later to observe the effect of each locally applied drug when compared to the control group (SRP plus water irrigation).

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic periodontitis with CAL ≥ 5 mm.
* No history of any systemic condition.
* Patient able to follow the required instructions.
* Willing to sign an informed consent form.
* Didn't receive any antibiotic therapy and periodontal therapy in the last 2-3 months.

Exclusion Criteria:

* Patients with systemic diseases that influence the condition (ex, hypertension, diabetes, kidney diseases and transplants).
* Patients who refuse to write an informed consent form.
* Smokers.
* Taking certain medications including antibiotics, antihypertensive, anticonvulsants, immunosuppressants, or any other drug that may affect the periodontal health status.
* Pregnant and lactating women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Measuring level of inflammatory markers MMP-9, TGF-Beta 1, IL-8, TIMP-1 in the gingival crevicular fluid | 14 days
  Level of selected inflammatory markers (MMP-9, TGF-Beta 1, IL-8, TIMP-1) is measured in the gingival crevicular fluid before and after use of different interventions
Measuring clinical attachment level | 14 days
  Clinical attachment level (CAL) is measured at baseline and after using different interventions
Measuring bleeding on probing | 14 day
  Measuring bleeding on probing (BOP), indicated by score 0 (no bleeding) score 1 (bleeding), from periodontal pockets treated with different interventions at baseline and at the end of the trial period.

CONTACTS AND LOCATIONS:
Overall Officials: Aya H Ali, Principal Investigator — College of Dentistry/ University of Baghdad
Locations (1):
- College of Dentistry/ University of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided